CLINICAL TRIAL: NCT00857493
Title: A Randomized, Double-blind, Placebo-controlled Phase II Study to Evaluate Safety and Immunogenicity of One and Two Doses of IMVAMUNE® Smallpox Vaccine in 56-80 Year Old Vaccinia-experienced Subjects
Brief Title: A Study to Evaluate Safety and Immunogenicity of One and Two Doses of IMVAMUNE® Smallpox Vaccine in 56-80 Year Old Vaccinia-experienced Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: POX-MVA-024
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental)
  Interventions: Biological: IMVAMUNE
- Group 2 (Experimental)
  Interventions: Biological: IMVAMUNE

INTERVENTIONS:
Biological: IMVAMUNE — Two s.c. vaccinations with 0.5 ml IMVAMUNE® vaccine containing 1 x 10E8 TCID50 / dose
  Arms: Group 1
Biological: IMVAMUNE — One s.c. vaccination with placebo (0.5 ml saline), followed by a second s.c. vaccination with 0.5 ml IMVAMUNE® vaccine containing 1 x 10E8 TCID50
  Arms: Group 2

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled Phase II Study to Evaluate Safety and Immunogenicity of One and Two Doses of IMVAMUNE® Smallpox Vaccine in 56-80 Year Old Vaccinia-Experienced Subjects

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 56-70 years of age. If no safety concerns are identified upon review of the safety data from the first 30 subjects enrolled, the age range is extended up to 80 years.
* Time since most current smallpox vaccination > 10 years.
* The subject has read, signed and dated the Informed Consent Form (ICF), successfully completed (at least 90% correct [no more than 3 attempts allowed]) the test of understanding and has signed the Health Insurance Portability and Accountability Act (HIPAA) authorization form.
* Women must have a negative serum pregnancy test at screening and negative urine pregnancy test within 24 hours prior to vaccination.
* Women of childbearing potential (WOCBP) must have used an acceptable method of contraception for 30 days prior to the first vaccination, must agree to use an acceptable method of contraception during the study and must not plan to become pregnant for at least 28 days after the last vaccination. (Acceptable contraception methods are restricted to abstinence, barrier contraceptives, intrauterine contraceptive devices or licensed hormonal products).
* Weight: ≥ 100 pounds (45.5 kg) and ≤ 330 pounds (150 kg).
* White blood cells ≥ 2500/mm3 and < 11,000/mm3.
* Absolute neutrophil count within normal limits.
* Hemoglobin within normal limits.
* Platelets within normal limits.
* Adequate renal function defined as:

  1. Urine protein ≤ +1 (by dip stick)
  2. Serum creatinine within normal limits
* Adequate hepatic function defined as:

  1. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) in the absence of other evidence of significant liver disease.
  2. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase ≤ 1.5 x ULN.
* Cardiac troponin I < 2 x ULN.
* Electrocardiogram (ECG) without clinically significant findings, e.g. any kind of atrioventricular or intraventricular conditions or blocks such as complete left or right bundle branch block, AV node block, QTc or PR prolongation, sustained atrial arrhythmias, sustained ventricular arrhythmia, 2 premature ventricular contractions (PVC) in a row, ST elevation consistent with ischemia.

Exclusion Criteria:

* History of or active immunodeficiency or immuno-suppression caused by acquired or congenital diseases or caused by treatments such as chronic administration (> 14 days) of systemic, i.e. parenteral or oral, corticosteroids (> 5 mg prednisone [or equivalent] per day), radiation or immune-modifying drugs.
* Periodic steroid injections, e.g. intraarticular, are not allowed within 30 days prior to the first vaccination and throughout the study until Visit 5 (V5).
* Post organ transplant subjects whether or not receiving chronic immunosuppressive therapy.
* Uncontrolled serious infection, i.e. not responding to antimicrobial therapy.
* History of any serious medical condition, which in the opinion of the investigator would compromise the safety of the subject or prevent the subject from complying with study requirements.
* History of or active autoimmune disease, e.g. Type I diabetes. Persons with vitiligo or thyroid disease taking thyroid hormone replacement are not excluded.
* Skin cancer in the past six months. If treatment for skin cancer was successfully completed more than six months ago and the malignancy is considered to be cured, the subject may be enrolled. Subjects with history of skin cancer must not be vaccinated at the previous site of cancer.
* Any other malignancy in the past five years. If treatment for cancer was successfully completed more than 5 years ago and the malignancy is considered to be cured, the subject may be enrolled.
* Clinically significant hematological, renal, hepatic, pulmonary, central nervous, cardiovascular or gastrointestinal disorders which are not adequately controlled by medical treatment within the last 12 weeks before vaccination as judged by the site's Principal Investigator.
* History of myocardial infarction, congestive heart failure with marked limitation of activity due to symptoms, e.g. walking short distances [20 100 m] (i.e. > Grade II according to the New York Heart Association), cardiomyopathy and stroke or transient ischemic attack in the past two years.
* Uncontrolled high blood pressure defined as systolic blood pressure ≥ 150 mm Hg and/or ≥ diastolic blood pressure ≥ 100 mm Hg within the last six months.
* Subjects with active coronary heart disease manifested by angina, even if on medication.
* 25 % or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's Risk Assessment Tool: http://hin.nhlbi.nih.gov/atpiii/calculator.asp
* Clinically significant mental disorder not adequately controlled by medical treatment.
* History of chronic alcohol abuse (40 g/day, e.g. 3 glasses of beer or 2 glasses of wine for at least six months) and/or intravenous drug abuse (within the last six months). Subjects with a history of other substance and/or alcohol abuse are also excluded if - in the opinion of the investigator - the abuse could prevent the subject from complying with study requirements.
* History of allergic disease or reactions likely to be exacerbated by IMVAMUNE® or any component of the vaccine, e.g. tris(hydroxymethyl)-amino methane, chicken embryo fibroblast proteins, aminoglycosides (gentamycin).
* History of anaphylactic shock or any severe allergic reaction to a vaccine requiring immediate treatment.
* Subjects undergoing treatment for tuberculosis infection or disease.
* Having received any vaccinations or planned vaccinations with a live vaccine within 30 days prior to or after study vaccination.
* Having received any vaccinations or planned vaccinations with a killed vaccine within 14 days prior to or after study vaccination.
* Administration or planned administration of immuno-globulins and/or any blood products during a period starting from three months prior to administration of the vaccine and ending at study conclusion.
* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned administration of such a drug during the study period.
* Temperature ≥ 100.4°F (38.0°C) at the time of enrollment.
* Any condition which might interfere with study objectives or would limit the subject's ability to complete the study in the opinion of the investigator.
* Study personnel.

Ages: 56 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard N Greenberg, MD, Principal Investigator — University of Kentucky
Locations (4):
- United States (4):
  - Orlando Clinical Research Center, Orlando, Florida
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, School of Medicine, Department of Medicine, Lexington, Kentucky
  - University of Rochester, Medical Center, Rochester, New York

REFERENCES:
- [Derived] Greenberg RN, Hay CM, Stapleton JT, Marbury TC, Wagner E, Kreitmeir E, Roesch S, von Krempelhuber A, Young P, Nichols R, Meyer TP, Schmidt D, Weigl J, Virgin G, Arndtz-Wiedemann N, Chaplin P. A Randomized, Double-Blind, Placebo-Controlled Phase II Trial Investigating the Safety and Immunogenicity of Modified Vaccinia Ankara Smallpox Vaccine (MVA-BN(R)) in 56-80-Year-Old Subjects. PLoS One. 2016 Jun 21;11(6):e0157335. doi: 10.1371/journal.pone.0157335. eCollection 2016. PMID 27327616

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 62 | 58
Completed (active study phase) | 59 | 58
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 62 | 58 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (5.41) | 62.6 (5.85) | 63.7 (5.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 40 | 77
  Male | 25 | 18 | 43

OUTCOME MEASURES:

1. Primary Outcome: Related Serious Adverse Events
Description: Incidence of Serious Adverse Events (SAEs) probably, possibly or definitely related to the trial vaccine
Time Frame: within 8 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 62 | 58
Participants | 0 | 0

2. Secondary Outcome: Unsolicited Non-serious AEs: Intensity
Description: Occurrence of unsolicited non-serious AEs by Intensity
Time Frame: within 29 days after any vaccination
Population: Safety Analysis Set
Measure: Number; unit: events
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 62 | 58
events
  Total | 73 | 58
  Grade 1 | 60 | 50
  Grade 2 | 9 | 7
  Grade 3 | 4 | 1
  Grade 4 | 0 | 0
  Missing | 0 | 0

3. Secondary Outcome: Unsolicited Non-serious AEs: Relationship to Vaccination
Description: Occurrence of unsolicited non-serious AEs by relationship to study vaccine
Time Frame: within 29 days after any vaccination
Population: Safety Analysis Set
Measure: Number; unit: events
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 62 | 58
events
  Unrelated/None | 32 | 26
  Unlikely | 6 | 2
  Possible | 20 | 13
  Probable | 8 | 5
  Definite | 7 | 12
  Missing | 0 | 0
  Total | 73 | 58

4. Secondary Outcome: Related Grade >=3 Adverse Events
Description: Incidence of any Grade >=3 Adverse Events probably, possibly or definitely related to the trial vaccine. Pooled solicited (general) and unsolicited AEs
Time Frame: within 29 days after any vaccination
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 62 | 58
Participants | 3 | 1

5. Secondary Outcome: Cardiac Signs or Symptoms
Description: Incidence, relationship and intensity of any cardiac sign or symptom indicating a case of myo-/pericarditis (AESI). AESIs were defined as any cardiac symptoms and ECG changes determined to be clinically significant or cardiac enzymes elevated above 2 x upper limit of normal range (ULN).
Time Frame: within 32 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 62 | 58
Participants
  Any AESI | 5 | 0
  Any AESI with intensity >= Grade 3 | 0 | 0
  Any AESI assessed as related to vaccine | 0 | 0

6. Secondary Outcome: Solicited Local Adverse Events
Description: Incidence and intensity of solicited local AEs (pain, erythema, swelling, induration, and pruritus). Percentages based on subjects with at least one completed diary card.
Time Frame: within 8 days after any vaccination
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 62 | 58
Participants
  Pain: Any | 46 | 36
  Pain: Grade >=3 | 4 | 1
  Erythema: Any | 49 | 37
  Erythema: Grade >=3 | 3 | 1
  Swelling: Any | 39 | 27
  Swelling: Grade >=3 | 0 | 0
  Induration: Any | 31 | 17
  Induration: Grade >=3 | 0 | 0
  Pruritis: Any | 27 | 22
  Pruritis: Grade >=3 | 0 | 0

7. Secondary Outcome: Solicited General Adverse Events
Description: Incidence of solicited general AEs (body temperature increased, headache, myalgia, chills, nausea, and fatigue): Intensity and relationship tovaccination. Percentages based on subjects with at least one completed diary card.
Time Frame: within 8 days after any vaccination
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 62 | 58
Participants
  Increased body temperature: Any | 2 | 1
  Increased body temperature: Related | 2 | 0
  Increased body temperature: Grade >=3 | 0 | 0
  Headache: Any | 19 | 22
  Headache: Related | 15 | 14
  Headache: Grade >=3 | 1 | 0
  Myalgia: Any | 19 | 14
  Myalgia: Related | 14 | 12
  Myalgia: Grade >=3 | 2 | 1
  Chills: Any | 5 | 4
  Chills: Related | 5 | 1
  Chills: Grade >=3 | 0 | 0
  Nausea: Any | 7 | 5
  Nausea: Related | 4 | 4
  Nausea: Grade >=3 | 0 | 0
  Fatigue: Any | 21 | 18
  Fatigue: Related | 18 | 15
  Fatigue: Grade >=3 | 1 | 0

8. Secondary Outcome: ELISA Response Rate
Description: Response rate based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Response is defined as the appearance of antibody titers ≥ detection limit (50) for initially seronegative subjects, or an increase of the antibody titer compared to Baseline titer for initially seropositive subjects. Individual peak response rate is based on the maximum post-Baseline antibody titer within 8 weeks (end of active trial phase). Percentages based on number of subjects with data available.
Time Frame: within 32 weeks
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 61 | 58
percentage of subjects
  Week 2 | 98.4 [91.2 to 100.0] | 19.0 [9.9 to 31.4]
  Week 4 | 96.6 [88.3 to 99.6] | 19.0 [9.9 to 31.4]
  Week 6 | 98.3 [91.1 to 100.0] | 96.6 [88.1 to 99.6]
  Week 8 | 100.0 [93.9 to 100.0] | 100.0 [93.8 to 100.0]
  Individual Peak | 100.0 [94.1 to 100.0] | 100.0 [93.8 to 100.0]
  Week 32 | 94.9 [85.9 to 98.9] | 82.8 [70.6 to 91.4]

9. Secondary Outcome: ELISA Seroconversion Rate
Description: Seroconversion rate based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Seroconversion is defined as the appearance of antibody titers ≥ detection limit (50) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Individual peak seroconversion rate is based on the maximum post-Baseline antibody titer within 8 weeks (end of active trial phase). Percentages based on number of subjects with data available.
Time Frame: within 32 weeks
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 61 | 58
percentage of subjects
  Week 2 | 83.6 [71.9 to 91.8] | 1.7 [0.0 to 9.2]
  Week 4 | 79.7 [67.2 to 89.0] | 3.4 [0.4 to 11.9]
  Week 6 | 83.3 [71.5 to 91.7] | 82.8 [70.6 to 91.4]
  Week 8 | 83.1 [71.0 to 91.6] | 77.6 [64.7 to 87.5]
  Individual Peak | 90.2 [79.8 to 96.3] | 84.5 [72.6 to 92.7]
  Week 32 | 59.3 [45.7 to 71.9] | 58.6 [44.9 to 71.4]

10. Secondary Outcome: ELISA GMT
Description: Geometric Mean Titers (GMT) based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Individual peak is defined as the maximum post-Baseline antibody titer within 8 weeks (end of active trial phase). Titers below the detection limit are included with a value of '1'.
Time Frame: within 32 weeks
Population: Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 61 | 58
Titer
  Week 0 | 129.0 [100.3 to 165.8] | 105.3 [71.8 to 154.5]
  Week 2 | 622.5 [491.2 to 788.9] | 98.5 [64.8 to 150.0]
  Week 4 | 501.2 [406.4 to 617.9] | 101.0 [66.5 to 153.3]
  Week 6 | 804.1 [636.3 to 1016.0] | 605.8 [479.6 to 765.2]
  Week 8 | 720.2 [577.9 to 897.6] | 505.0 [398.2 to 640.3]
  Individual Peak | 992.4 [769.2 to 1280.3] | 645.2 [505.0 to 824.3]
  Week 32 | 344.6 [288.9 to 411.1] | 258.1 [202.5 to 328.9]

11. Secondary Outcome: PRNT Response Rate
Description: Response rate based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT). Response is defined as the appearance of antibody titers ≥ detection limit (15) for initially seronegative subjects, or an increase of the antibody titer compared to Baseline titer for initially seropositive subjects. Individual peak response rate is based on the maximum post-Baseline antibody titer within 8 weeks (end of active trial phase). Percentages based on number of subjects with data available.
Time Frame: within 32 weeks
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 61 | 58
percentage of subjects
  Week 2 | 83.6 [71.9 to 91.8] | 15.5 [7.3 to 27.4]
  Week 4 | 81.4 [69.1 to 90.3] | 10.3 [3.9 to 21.2]
  Week 6 | 96.7 [88.5 to 99.6] | 82.8 [70.6 to 91.4]
  Week 8 | 89.8 [79.2 to 96.2] | 79.3 [66.6 to 88.8]
  Individual Peak | 96.7 [88.7 to 99.6] | 84.5 [72.6 to 92.7]
  Week 32 | 66.1 [52.6 to 77.9] | 50.0 [36.6 to 63.4]

12. Secondary Outcome: PRNT Seroconversion Rate
Description: Seroconversion rate based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT). Seroconversion is defined as the appearance of antibody titers ≥ detection limit (15) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Individual peak seroconversion rate is based on the maximum post-Baseline antibody titer within 8 weeks (end of active trial phase). Percentages based on number of subjects with data available.
Time Frame: within 32 weeks
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 61 | 58
percentage of subjects
  Week 2 | 73.8 [60.9 to 84.2] | 10.3 [3.9 to 21.2]
  Week 4 | 71.2 [57.9 to 82.2] | 8.6 [2.9 to 19.0]
  Week 6 | 90.0 [79.5 to 96.2] | 77.6 [64.7 to 87.5]
  Week 8 | 86.4 [75.0 to 94.0] | 74.1 [61.0 to 84.7]
  Individual Peak | 95.1 [86.3 to 99.0] | 77.6 [64.7 to 87.5]
  Week 32 | 55.9 [42.4 to 68.8] | 41.4 [28.6 to 55.1]

13. Secondary Outcome: PRNT GMT
Description: Geometric Mean Titers (GMT) based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT). Individual peak is defined as the maximum post-Baseline antibody titer within 8 weeks (end of active trial phase). Titers below the detection limit are included with a value of '1'.
Time Frame: within 32 weeks
Population: Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 61 | 58
Titer
  Week 0 | 11.9 [7.4 to 19.1] | 11.3 [6.5 to 19.4]
  Week 2 | 111.4 [72.0 to 172.2] | 9.2 [5.3 to 15.8]
  Week 4 | 79.5 [52.1 to 121.3] | 11.3 [6.8 to 18.7]
  Week 6 | 210.3 [146.1 to 302.7] | 126.7 [82.4 to 194.8]
  Week 8 | 144.9 [96.1 to 218.6] | 99.5 [63.8 to 155.1]
  Individual Peak | 257.6 [178.6 to 371.5] | 139.6 [89.2 to 218.5]
  Week 32 | 47.0 [31.1 to 71.1] | 27.6 [17.0 to 44.8]

14. Secondary Outcome: Correlation PRNT vs ELISA Titers
Description: Pearson Correlation Coefficient between the log10 transformed PRNT titers and the log10 transformed ELISA titers
Time Frame: within 32 weeks
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Pearson correlation coefficient
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 61 | 58
Pearson correlation coefficient
  Week 2 | 0.704 [0.546 to 0.810] | 0.489 [0.261 to 0.661]
  Week 4 | 0.569 [0.362 to 0.718] | 0.492 [0.264 to 0.664]
  Week 6 | 0.660 [0.484 to 0.781] | 0.697 [0.531 to 0.808]
  Week 8 | 0.600 [0.402 to 0.740] | 0.616 [0.421 to 0.752]
  Week 32 | 0.500 [0.276 to 0.668] | 0.654 [0.472 to 0.778]

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/58
Serious Adverse Events (participants affected / at risk) | 2/62 | 2/58
Other Adverse Events (participants affected / at risk) | 21/62 | 21/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=62) | Group 2 (N=58)
Cellulitis (Infections and infestations) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=62) | Group 2 (N=58)
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Application site haematoma (General disorders) | 0 | 3
Injection site haematoma (General disorders) | 1 | 5
Injection site nodule (General disorders) | 4 | 2
Injection site pain (General disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1
Lymphocyte count decreased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes